CLINICAL TRIAL: NCT01254773
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center, Biomarker, Safety, and Pharmacokinetic Study of Bapineuzumab (AAB-001) Administered Subcutaneously at Monthly Intervals in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Amyloid Imaging And Safety Study Of Subcutaneous Bapineuzumab In Subjects With Mild to Moderate Alzheimer's Disease
Acronym: SUMMIT AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAB-001-SC-ALZ-2003
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bapineuzumab SC Dose 1; 2 mg (Experimental)
  Interventions: Drug: Experimental Bapineuzumab
- Bapineuzumab SC Dose 2; 7 mg (Experimental)
  Interventions: Drug: Experimental Bapineuzumab
- Bapineuzumab SC Dose 3; 20 mg (Experimental)
  Interventions: Drug: Experimental Bapineuzumab
- Placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Experimental Bapineuzumab — Bapineuzumab 2 mg, Bapineuzumab 7 mg, Bapineuzumab 20 mg, Placebo
  Arms: Bapineuzumab SC Dose 1; 2 mg; Bapineuzumab SC Dose 2; 7 mg; Bapineuzumab SC Dose 3; 20 mg

SUMMARY:
This study in individuals with mild to moderate Alzheimer's Disease is designed to assess:(1) safety and tolerability (2) the capacity of subcutaneous bapineuzumab to reduce brain amyloid load as measured by positron emission tomography (PET) scans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Age from 50 to less than 89
* Mini-Mental Status Exam score of 18-26 inclusive
* Brain magnetic resonance imaging (MRI) scan consistent with the diagnosis of AD
* Stable doses of medications (cholinesterase inhibitors and memantine allowed)
* Caregiver able to attend all clinic visits with patient
* Amyloid burden on screening PET scan consistent with diagnosis of AD

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Significant systemic illness
* History of stroke or seizure, autoimmune disease, myocardial infarction within the last 2 years
* Smoking greater than 20 cigarettes per day
* Anticonvulsants, anti-Parkinson's, anticoagulant, or narcotic medications
* Prior treatment experimental immunotherapeutics or vaccines for AD
* Women of childbearing potential
* Presence of pacemakers, CSF shunts, or foreign metal objects in the eyes, skin or body

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of bapineuzumab administered subcutaneously (SC) at monthly intervals compared to placebo on cerebral amyloid burden in subjects with mild to moderate AD. | 24 months

SECONDARY OUTCOMES:
To assess the safety of bapineuzumab administered SC at monthly intervals compared to placebo in subjects with mild to moderate AD | 24 months
To assess the effect of bapineuzumab administered SC at monthly intervals compared to placebo on cognitive and functional endpoints. | 24 months

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Janssen AI Investigational Site, Tucson, Arizona
  - Janssen AI Investigational Site, La Habra, California
  - Janssen AI Investigational Site, Lomita, California
  - Janssen AI Investigational Site, Long Beach, California
  - Janssen AI Investigational Site, Oceanside, California
  - Janssen AI Investigational Site, Pasadena, California
  - Janssen AI Investigational Site, Santa Monica, California
  - Janssen AI Investigational Site, Sherman Oaks, California
  - Janssen AI Investigational Site, Deerfield Beach, Florida
  - Janssen AI Investigational Site, Delray Beach, Florida
  - Janssen AI Investigational Site, Fort Meyers, Florida
  - Janssen AI Investigational Site, Miami Springs, Florida
  - Janssen AI Investigational Site, South Miami, Florida
  - Janssen AI Investigational Site, Atlanta, Georgia
  - Janssen AI Investigational Site, Indianapolis, Indiana
  - Janssen AI Investigational Site, Kansas City, Kansas
  - Janssen AI Investigational Site, Lexington, Kentucky
  - Janssen AI Investigational Site, Plymouth, Massachusetts
  - Janssen AI Investigational Site, Farmington Hills, Michigan
  - Janssen AI Investigational Site, Creve Coeur, Missouri
  - Janssen AI Investigational Site, St Louis, Missouri
  - Janssen AI Investigational Site, Latham, New York
  - Janssen AI Investigational Site, Winston-Salem, North Carolina
  - Janssen AI Investigational Site, Dayton, Ohio
  - Janssen AI Investigational Site, Portland, Oregon
  - Janssen AI Investigational Site, Philadelphia, Pennsylvania
  - Janssen AI Investigational Site, Providence, Rhode Island